CLINICAL TRIAL: NCT04544566
Title: A Clinical Pilot Study of Newly Developed Ostomy Tapes and How They Adhere to the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP319
Record Dates: First submitted 2020-06-26; First posted 2020-09-10 (Actual); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Stoma Site Leakage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product A new adhesive material (Experimental): The adhesives in the ostomy tapes are developed to make the tape seal to the skin and thereby minimise the risk of leakage episodes. At the same time, the tape should be easy to remove without affecting the skin.
  Interventions: Device: Test product A; Device: Test product B; Device: Comparator
- Test product B new adhesion material (Experimental): The adhesives in the ostomy tapes are developed to make the tape seal to the skin and thereby minimise the risk of leakage episodes. At the same time, the tape should be easy to remove without affecting the skin.
  Interventions: Device: Test product A; Device: Test product B; Device: Comparator
- Comparator (Active Comparator): The comparator product is Brava Elastic tape which is already on the market and will be used within the in-tended use in this clinical investigation.
  Interventions: Device: Test product A; Device: Test product B; Device: Comparator

INTERVENTIONS:
Device: Test product A — one new adhesive material which is applied to the baseplate and the subjects peristomal skin
Device: Test product B — one new adhesive material which is applied to the baseplate and the subjects peristomal skin
Device: Comparator — Already CE- marked product as a comparator which is applied to the baseplate and the subjects peristomal skin

SUMMARY:
An investigation of non-CE marked stoma tape products. This investigation is a randomised, open-label, comparative, cross-over study, with three test periods. In total, 12 subjects will be included and randomised.

DETAILED DESCRIPTION:
The test products are non-CE marked stoma tape products. This investigation is a randomised, open-label, comparative, cross-over study, with three test periods. In total, 12 subjects will be included and randomised.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent
* Be at least 18 years of age and have full legal capacity
* Have had a stoma for more than ½ year
* Have intact skin on the area used in the study (Assessed by investigator, see Appendix 1).
* Willing to change baseplate every second day or less frequent
* Willing to avoid using Concave baseplate during the study.
* Willing to avoid the use of barrier creams or similar that affect the skin/adhesive interface under the tape.

Exclusion Criteria:

* Currently receiving or have within the past 2 months received radio-and/or chemotherapy
* Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet(injection) treatment
* Is pregnant or breastfeeding
* Having dermatological problems in the peristomal area (assessed by investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Karlsmark, MD, Principal Investigator — Bispebjerg hospital, Dermato-Venerologisk afdeling.
Locations (1):
- Bispebjerg hospital, Copenhagen, Copenhagen NV, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects that met the inclusion and exclusion criteria was randomised to one of six treatment arms. Each arm examined the Comparator Tape and the two Test Tapes in various orders.
Groups:
- Test Tape A, Test Tape B, and Then Comparator Tape; Test Tape A, Comparator Tape and Then Test Tape B; Comparator Tape, Test Tape A and Then Test Tape B; Comparator Tape, Test Tape B and Then Test Tape A; Test Tape B, Comparator Tape and Then Test Tape A; Test Tape B, Test Tape A and Then Comparator Tape: The adhesives in the ostomy tapes are developed to make the tape seal to the skin and thereby minimise the risk of leakage episodes. At the same time, the tape should be easy to remove without affecting the skin.
  Test product A: one new adhesive material was applied to the baseplate and the subjects peristomal skin
  Test product B: one new adhesive material was applied to the baseplate and the subjects peristomal skin.
  The comparator product is Brava Elastic tape which is a CE marked product already on the market and applied to the baseplate and the subjects peristomal skin. The product was used within the in-tended use in this clinical investigation.
Period: Overall Study
Arm/Group | Test Tape A, Test Tape B, and Then Comparator Tape | Test Tape A, Comparator Tape and Then Test Tape B | Comparator Tape, Test Tape A and Then Test Tape B | Comparator Tape, Test Tape B and Then Test Tape A | Test Tape B, Comparator Tape and Then Test Tape A | Test Tape B, Test Tape A and Then Comparator Tape
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject from treatment arm 6 did not complete the questionnaires related to secondary endpoints
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Tape A, Test Tape B, and Then Comparator Tape | Test Tape A, Comparator Tape and Then Test Tape B | Comparator Tape, Test Tape A and Then Test Tape B | Comparator Tape, Test Tape B and Then Test Tape A | Test Tape B, Comparator Tape and Then Test Tape A | Test Tape B, Test Tape A and Then Comparator Tape | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 2 | 1 | 0 | 4
  >=65 years | 1 | 2 | 2 | 0 | 1 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (26.2) | 71 (0) | 71.5 (6.4) | 42.5 (30.4) | 63 (19.8) | 66 (0) | 61.1 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 2 | 2 | 6
  Male | 1 | 2 | 2 | 1 | 0 | 0 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 2 | 2 | 2 | 2 | 2 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Adherent Area Measured by Photo of Used Tape
Description: The adherent area (cm2) measured per baseplate change after use shows how effectively the ostomy tape adheres to the skin. After removal of the ostomy tape, a photo of the tape was taken. The adherent area was measured from the photo and an image analysing program.
Time Frame: Tapestrips per test product were removed from the baseplate at each product change and saved for the next site visit every 7-9 days for evaluation
Measure: Least Squares Mean (Standard Deviation); unit: Cm2
Groups:
- Comparator: The comparator product is Brava Elastic tape which is already on the market and will be used within the intended use in this clinical investigation.
  Test product A: one new adhesive material which is applied to the baseplate and the subjects peristomal skin
  Test product B: one new adhesive material which is applied to the baseplate and the subjects peristomal skin
  Comparator: Already CE- marked product as a comparator which is applied to the baseplate and the subjects peristomal skin
Arm/Group | Test Product A New Adhesive Material | Test Product B New Adhesion Material | Comparator
Number analyzed (Participants) | 12 | 12 | 12
Cm2 | 46.54 (1.23) | 51.61 (1.24) | 52.94 (1.24)

2. Secondary Outcome: Erythema Measured After Each Treatment Period by Spectrophotometric Method
Description: A change in the surface skin colour is known to be related to a change in the blood flow. This can be measured non-invasively with a spectrophotometric instrument (Derma-spectrophotometer, Cortex Technology A/S, Hadsund) where redness of the skin is measured. The measurement of erythema is based on an active color detecting chip. Illumination is provided by two high intensity white LEDs. The spectrophotometer accommodates the color sensor, filters, optics and light source. Light is provided by two high intensity with LEDs and a unique feature is the guiding light, which illuminates the target during the positioning of the device. The LEDs illuminates the target area and the skin color measurement is performed. The measurements performed with the spectrophotometric instrument do not have units. But the measures are used for the estimation of the level of the redness (hemoglobin) in the skin. The higher the value, the more pigment in the skin.
Time Frame: The measurements were carried out after 7-9 days of treatment with the test tape
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Test Product A New Adhesive Material | Test Product B New Adhesion Material | Comparator
Number analyzed (Participants) | 12 | 12 | 12
Unitless | 10.1 (2.6) | 10.0 (3.0) | 11.0 (3.7)

3. Secondary Outcome: Erythema Measured After Tape Removal by Photos
Description: A change in the surface skin colour is known to be related to a change in the blood flow. This can be measured non-invasively with a spectrophotometric instrument (Derma-spectrophotometer, Cortex Technology A/S, Hadsund) where both the redness and the colour of the skin are measured. Furthermore, visual assessments of photos have been used in several exploratory clinical investigations by Coloplast A/S to explore how adhesives affect the skin. The visual assessment is conducted by trained personnel and is a valuable tool for assessing newly developed adhesives and their impact on skin in the early development phases.
Time Frame: The measurements were carried out after 7-9 days of treatment with the test tape
Population: One subject from treatment-arm 6 is missing from the analysis as the photo material of the subject was insufficient for assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product A New Adhesive Material | Test Product B New Adhesion Material | Comparator
Number analyzed (Participants) | 11 | 11 | 11
Participants
  Lowest degree of skin reaction | 6 | 6 | 3
  Middle degree of skin reaction | 1 | 4 | 2
  Highest degree of skin reaction | 4 | 1 | 6

4. Secondary Outcome: Feeling of Security
Description: Subjects will be asked how they rate feeling of security ("How was the feeling of security?) on a five point scale, when wearing the tape; 1. Very Poor, 2. Poor, 3. Acceptable, 4. Good, 5. Very Good.
Time Frame: The evaluation was carried out after 7-9 days of treatment with the test tape
Measure: Count of Units; unit: Product change
Units Other Than Participants: Product change
Arm/Group | Test Product A New Adhesive Material | Test Product B New Adhesion Material | Comparator
Number analyzed (Participants) | 11 | 11 | 11
Number analyzed (Product change) | 52 | 49 | 47
Product change
  Very poor | 3 | 0 | 0
  Poor | 9 | 0 | 0
  Acceptable | 14 | 2 | 4
  Good | 15 | 25 | 14
  Very good | 11 | 22 | 29

5. Secondary Outcome: Adhesion of Tape
Description: Subjects will be asked how they perceive the immediate adhesion to the skin ("how was the immediate adhesion to the skin?) and rate adhesion on a five-point scale: 1. Very poor, 2. Poor, 3. Acceptable, 4. Good, 5. Very good.
Time Frame: The evaluation was carried out after 7-9 days of treatment with the test tape
Measure: Count of Units; unit: Product change
Units Other Than Participants: Product change
Arm/Group | Test Product A New Adhesive Material | Test Product B New Adhesion Material | Comparator
Number analyzed (Participants) | 11 | 11 | 11
Number analyzed (Product change) | 52 | 49 | 47
Product change
  Very poor | 5 | 0 | 0
  Poor | 11 | 0 | 0
  Acceptable | 16 | 6 | 1
  Good | 12 | 22 | 9
  Very good | 8 | 21 | 37

6. Secondary Outcome: Comfort
Description: Subjects will be asked how they perceived the comfort of the tape ("How comfortable was the tape to wear?") and rate comfort on a 5-pont scale; 1. very discomfortable, 2. Discomfortable, 3. Acceptable, 4. Comfortable, 5. Very comfortable.
Time Frame: The evaluation was carried out after 7-9 days of treatment with the test tape
Measure: Count of Units; unit: Product change
Units Other Than Participants: Product change
Arm/Group | Test Product A New Adhesive Material | Test Product B New Adhesion Material | Comparator
Number analyzed (Participants) | 11 | 11 | 11
Number analyzed (Product change) | 52 | 49 | 47
Product change
  Very discomfortable | 2 | 3 | 0
  Discomfortable | 5 | 5 | 2
  Acceptable | 14 | 2 | 3
  Comfortable | 19 | 24 | 21
  Very comfortable | 12 | 15 | 21

7. Secondary Outcome: Skin Issues in the Area Covered by the Tape
Description: Subjects will be asked if they had any skin-related complications in the area covered by the tape (yes, no).
Time Frame: The evaluation was carried out after 7-9 days of treatment with the test tape
Measure: Count of Units; unit: Product change
Units Other Than Participants: Product change
Arm/Group | Test Product A New Adhesive Material | Test Product B New Adhesion Material | Comparator
Number analyzed (Participants) | 11 | 11 | 11
Number analyzed (Product change) | 52 | 49 | 47
Product change
  Complications where tape was applied - Yes | 18 | 13 | 6
  Complications were tape was applied- No | 34 | 36 | 41

8. Secondary Outcome: Adverse Events
Description: All Adverse Events are captured and documented throughout the study.
Time Frame: 27 days
Measure: Count of Participants; unit: Participants
Groups:
- Test Tape A: The adhesives in the ostomy tapes are developed to make the tape seal to the skin and thereby minimise the risk of leakage episodes. At the same time, the tape should be easy to remove without affecting the skin.
  Test product A: one new adhesive material was applied to the baseplate and the subjects peristomal skin
- Test Tape B: The adhesives in the ostomy tapes are developed to make the tape seal to the skin and thereby minimise the risk of leakage episodes. At the same time, the tape should be easy to remove without affecting the skin.
  Test product B: one new adhesive material was applied to the baseplate and the subjects peristomal skin.
- Comparator Tape: The adhesives in the ostomy tapes are developed to make the tape seal to the skin and thereby minimise the risk of leakage episodes. At the same time, the tape should be easy to remove without affecting the skin.
  The comparator product is Brava Elastic tape which is a CE marked product already on the market and applied to the baseplate and the subjects peristomal skin. The product was used within the intended use in this clinical investigation.
Arm/Group | Test Tape A | Test Tape B | Comparator Tape
Number analyzed (Participants) | 12 | 12 | 12
Participants | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study period for a maximum of 27 days. If subject had on-going SAEs at termination, they were followed until the event was solved or until the subject could no longer be followed (lost to follow up). Subjects without SAEs or with terminated SAEs were not followed-up upon after the final termination visit.
Arm/Group | Test Product A New Adhesive Material | Test Product B New Adhesion Material | Comparator
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product A New Adhesive Material (N=12) | Test Product B New Adhesion Material (N=12) | Comparator (N=12)
Non serious adverse event (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Erosion of peristomal skin
Non serious adverse event (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Parodontitis Spicalis

LIMITATIONS AND CAVEATS:
One subject missed completing questionnaire related to secondary end points for Test Tape A and Comparator Tape and one subject was included in the study despite treatment with steroid cream of pyoderma ulcers. The treatment was close to being completed and was assessed by investigator as a deviation that had no impact on the rights, safety and well-being of the subject or that could impact the scientific outcome of the investigation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT04544566/Prot_SAP_000.pdf